CLINICAL TRIAL: NCT03733847
Title: Rehabilitation Trajectories. A Study of Rehabilitation Processes Across Health Care Levels in Patients With Rheumatic and Musculoskeletal Diseases
Brief Title: Rehabilitation Trajectories
Status: Completed | Type: Observational
Sponsor: National Resource Center for Rehabilitation in Rheumatology (Other)
Collaborators: Haugesund Rheumatism Hosptial AS (Unknown); Betanien Hospital (Other); Vikersund Rehabilitation Center AS (Unknown); Meråker Rehabilitation Center (Unknown); North Norway Rehabilitation Center (Other); UniCare Jeløy (Unknown); Sørlandet Hospital (Unknown); Innlandet HF Konsvinger Hospital (Unknown); Rehab Vest Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, Ingvild Kjeken, Professor, National Resource Center for Rehabilitation in Rheumatology
Other Study IDs: Project nr. 97035
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Musculoskeletal Disease
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this multicentre cohort study is to provide evidence that can be used to improve continuity and quality in rehabilitation practice and rehabilitation processes across health care levels for patients with rheumatic and musculoskeletal diseases (RMDs).

DETAILED DESCRIPTION:
There is an urgent need to develop rehabilitation trajectories that ensure coordination and communication between health care levels, support of self-management and self-monitoring, and follow-up tailored to patients' needs. Such trajectories should be based on evidence from current practice. The "Rehabilitation trajectories" project will systematically explore and describe current practice of planned and implemented follow-up and self-management strategies in primary health care during the first year after rehabilitation for patients with musculoskeletal diseases. Further, a newly developed core set of PROMs designed for evaluation of rehabilitation in RMDs and a self-monitoring web-based system will be tested for feasibility. Knowledge of patients' experiences and use of this self-monitoring system as a self-management and communication tool is needed in order to improve and integrate such e-technology in future care.

The Rehabilitation Trajectory study is a multi-centre study, led by the National Unit on Rehabilitation in Rheumatology and including participants at four rheumatology hospital departments and five specialized rehabilitation institutions. Participants will thus be included from all four health regions in Norway.

The study has five points of assessment. In an electronic portal, delivered by CheckWare, patients will log in with their Bank ID and complete the core set of PROMs at admission, discharge, and 4, 8 and 12 months following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to rehabilitation at one of the nine participating rehabilitation centres with one of the following groups of diagnosis: Inflammatory rheumatic disease, Osteoarthritis, Low back pain, Neck/shoulder pain, Generalized pain syndromes (including fibromyalgia), Osteoporosis, Connective tissue diseases (SLE, Lupus, Myositis etc.), Fractures with need of rehabilitation, or Rehabilitation after orthopaedic surgery. Good proficiency in oral and written Norwegian language. Access to internet and BankID.

Exclusion Criteria:

* Cognitive impairment or severe mental illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatic and musculoskeletal diseases from Norway admitted to rehabilitation at one of the nine participating rehabilitation centres.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Goal attainment | One year
  Goal attainment will be measures by the Patient Specific Functional Scale. Scale from 0 to 10, were 10 is the best score. Mean score is calculated from all activites scored.

SECONDARY OUTCOMES:
Health-realted quality of life | One year
  Health-realted quality of life will be measured by the EQ5D
Physical function | One year
  Physical function will be measured by the 30 seconds sit to stand test

OTHER OUTCOMES:
General Pain | One year
  Pain will be measured on a numeric rating scale (NRS). Pain is measured on a subjective scale from 0 to 10, were 0 is no pain and 10 is the worst pain.
Fatigue | One year
  Fatigue will be measured on a numeric rating scale (NRS). Fatigue is measured on a subjective scale from 0 to 10, were 0 is no fatiuge and 10 is the worst abount of fatigue.
Motivation for goal attainment | One year
  Motivation for goal attainment will be measured on a numeric rating scale (NRS). Motivation is measured on a subjective scale from 0 to 10, were 0 is no motviation and 10 is the best and highest motivation.
Function in daily acitvities | One year
  Daily activities will be measured by the Hannover Functional Ability Questionnair
Coping | One year
  Coping will be measures by the Effective Musculoskeletal Consumer Scale. The scale goes from 0 to 4, were 0 stated "never" and 4 states "always".
Mental health | One year
  Mental health will be measured by the Hopkins Symptoms Checklist
Participation | One year
  Participation will be measured by the participation scale in COOP/WONKA

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, PhD, Study Director — Diakonhjemmet Hospital